CLINICAL TRIAL: NCT02017015
Title: A PHASE 2, MULTI-CENTER STUDY TO EVALUATE THE SAFETY AND EFFICACY OF ABI-007 PLUS GEMCITABINE IN CHINESE PATEINTS WITH METASTATIC PANCREATIC ADENOCARCINOMA
Brief Title: Safety and Efficacy Study of Nab-paclitaxel Plus Gemcitabine in Chinese Patients With Metastatic Pancreatic Cancer
Acronym: PANC-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABI-007-PANC-001
Record Dates: First submitted 2013-12-05; First posted 2013-12-20 (Estimated); Results first posted 2016-11-22 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic cancer; Metastatic pancreatic cancer; treatment for pancreatic cancer; Abraxane clinical research trials; Celgene clinical research trials
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- nab-paclitaxel with gemcitabine (Experimental): nab-paclitaxel at 125 mg/m^2, intravenous (IV) infusion over 30 to 40 minutes followed by gemcitabine at 1000 mg/ m^2 IV infusion over 30 to 40 minutes given once weekly for 3 weeks (Days 1, 8 and 15) followed by a week of rest (28 day cycle).
  Interventions: Drug: nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: nab-paclitaxel — nab-paclitaxel at 125 mg/m^2, by IV infusion over 30 to 40 minutes (maximum infusion time not to exceed 40 minutes)
  Other Names: ABI-007; Abraxane
Drug: Gemcitabine — Gemcitabine at 1000 mg/m^2 IV infusion over 30 to 40 minutes given once weekly for 3 weeks (Days 1, 8 and 15) followed by a week of rest (28 day cycle).
  Other Names: Gemzar

SUMMARY:
The purpose of this study is to determine the safety and efficacy of nab-paclitaxel combined with gemcitabine in Chinese patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This is a Phase 2 trial in China to evaluate the safety and efficacy of the combination of nab-paclitaxel and gemcitabine administered in patients diagnosed with metastatic pancreatic adenocarcinoma. This study is designed to be a Chinese bridging study to complement the Global pivotal study (CA-046).

The study consists of three parts: (1) Dose evaluation; (2) Single arm to evaluate efficacy following an optimal Simon two-stage design; and (3) Randomized 2-arm to evaluate the efficacy and safety of nab-paclitaxel plus gemcitabine versus gemcitabine alone. These 3 parts will be carried out sequentially. The Part 3 randomized 2-arm portion will only be carried out if deemed necessary per protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has definitive histologically or cytologically confirmed metastatic pancreatic adenocarcinoma (Islet cell neoplasms are excluded) that is measurable by Response Evaluation criteria for solid tumors (RECIST V1.0)
2. Patients must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic pancreatic cancer. Prior treatment with 5-fluorouracil (5-FU) or gemcitabine administered as a radiation sensitizer in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present. Patients having received cytotoxic doses of gemcitabine or any other chemotherapy in the adjuvant setting are not eligible for this study
3. Patient has a Karnofsky performance status (KPS) ≥ 70
4. Initial diagnosis of metastatic disease must have occurred ≤ 6 weeks prior to starting Cycle 1 Day 1. NOTE: the clock for this time interval starts with the date of last evaluation confirming pancreatic metastatic disease (either biopsy or imaging results)
5. Patients should be asymptomatic for jaundice prior to Cycle 1 Day 1. Significant or symptomatic amounts of ascites should be drained prior to Cycle 1 Day 1. Pain symptoms should be stable and should not require modifications in analgesic management prior to Cycle 1 Day 1
6. Patient has adequate blood counts at screening (obtained ≤ 14 days prior to starting Cycle 1 Day 1):

   * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
   * Platelet count ≥ 100,000/mm^3 (100 × 10^9/L);
   * Hemoglobin (Hgb) ≥ 9 g/dL
7. Patient has the following blood chemistry levels at Screening (obtained ≤ 14 days prior to starting Cycle 1 Day 1):

   * Aspartate aminotransferase (SGOT) and alanine transaminase (SGPT) are ≤ 2.5 upper limit of normal (ULN) range, unless liver metastases are clearly present, then ≤ 5 × upper limit of normal (ULN) range is allowed
   * Total bilirubin ≤ upper limit of normal range
   * Serum creatinine within normal limits or calculated clearance ≥ 60 mL/min/1.73 m^2 for patients with serum creatinine levels above or below the institutional normal value. If using creatinine clearance, actual body weight should be used for calculating creatinine clearance (eg, using the Cockcroft-Gault formula). For patients with a body mass index (BMI) > 30 kg/m^2, lean body weight should be used instead.
8. The patient has acceptable coagulation studies (obtained ≤14 days prior to starting Cycle 1 Day 1) as demonstrated by prothrombin time (PT) and partial thromboplastin time (PTT) within normal limits (WNL) ±15%.
9. The patient has no clinically significant abnormalities in urinalysis results (obtained ≤14 days prior to starting Cycle 1 Day 1).
10. Male or non-pregnant and non-lactating female, and ≥ 18 years of age at the time of signing the informed consent document.

    * If a female patient is of child-bearing potential, as evidenced by regular menstrual periods, she must have a negative pregnancy test (e.g. serum β-subunit of human chorionic gonadotropin (β-hCG) documented prior to the first administration of study drug.
    * If sexually active, the patient must agree to use contraception considered adequate and appropriate by the Investigator during the period of administration of study drug. In addition, male and female patients must utilize contraception after the end of treatment as recommended in the product's
11. Patient has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent Form prior to participation in any study-related activities.
12. Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Patient has known brain metastases
2. Patient has only locally advanced disease.
3. Patient has a ≥ 20% decrease in serum albumin level between Screening visit and within 72 hours prior to Cycle 1 Day 1.
4. History of malignancy in the last 5 years (including chronic leukemias). Patients with prior history of in situ cancer or basal or squamous cell skin cancer are eligible. Patients with other malignancies are eligible if they were cured by surgery alone or surgery plus radiotherapy and have been continuously disease-free for at least 5 years.
5. Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
6. Patient has known infection with human immunodeficiency virus, and/or active infection with hepatitis B, or hepatitis C (patients with known historical infection with hepatitis B or C should be discussed with the Sponsor).
7. Patient has undergone major surgery, other than diagnostic surgery (ie, surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.
8. Patient that has a history of a myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) Class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or electrocardiogram (ECG) abnormality, cerebrovascular accident, transient ischemic attack, seizure disorder or clinically significant cardiac dysrhythmia or ECG abnormality, within 6 months prior to Cycle 1 Day 1
9. Patient has a history of allergy or hypersensitivity to any of the study drugs or any of their excipients, or the patient exhibits any of the adverse events .
10. History of connective tissue disorders (eg, lupus, scleroderma, arteritis nodosa).
11. Patients with a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies.
12. Patient has any condition, including serious medical risk factors, medical conditions, laboratory abnormalities or psychiatric disorders, which could compromise the patient's safety or the study data integrity.
13. Patient is enrolled in any other clinical protocol or investigational trial with an interventional agent or assessments that may interfere with study procedures.
14. Patient is unwilling or unable to comply with study procedures, or is planning to take vacation for 7 or more consecutive days during the treatment phase of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2013-12-24 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2016-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lu, MD, Study Director — Celgene
Locations (15):
- China (15):
  - 307 Hospital of Chinese PLA, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Beijing Cancer Hospital, Beijing, PR
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang
  - Harbin Medical University Tumor Hospital, Harbin, Heilongjiang
  - Jiangsu Province Hospital The First Hospital affiliated with Nanjing Medical University, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Xijing Hospital, Xi'an
  - Henan Cancer Hospital, Zhengzhou

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multi-center study was conducted by investigators in China and enrolled patients at a total of 13 sites. This study was designed to be a Chinese bridging study to complement the global pivotal study (CA046).
Groups:
- Nab-paclitaxel and Gemcitabine: Nab-paclitaxel 125 mg/m^2 by intravenous (IV) infusion over 30 - 40 minutes followed by gemcitabine 1000 mg/ m^2 by IV infusion over 30 - 40 minutes once weekly for 3 weeks (Days 1, 8 and 15) followed by one week of rest (28 day cycle).
Period: Overall Study
Arm/Group | Nab-paclitaxel and Gemcitabine
Started | 83
Safety Population | 83
Completed | 14 (Completed = Participants remaining on treatment at the time of the data cut-off of 01 Jun 2015)
Not Completed | 69
Not completed — Adverse Event | 9
Not completed — Withdrawal by Subject | 21
Not completed — Death | 4
Not completed — Progressive Disease | 31
Not completed — Non-compliance with study drug | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population includes all enrolled participants
Groups:
- Nab-paclitaxel and Gemcitabine: Nab-paclitaxel 125 mg/m^2 by intravenous (IV) infusion over 30 - 40 minutes followed by gemcitabine 1000 mg/ m2 IV infusion over 30 - 40 minutes once weekly for 3 weeks (Days 1, 8 and 15) followed by one week of rest (28 day cycle).
Arm/Group | Nab-paclitaxel and Gemcitabine
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 58
Region of Enrollment [Number; unit: participants]
  China | 83
Karnofsky Performance Status (KPS) [Number; unit: participants] — The Karnofsky Performance Status Scale (KPS) was designed to measure the level of participant activity and medical care requirements. A general measure of participant independence and has been widely used as a general assessment of participants with cancer. The Karnofsky score runs from 100 to 0, where 100 is "perfect" health and 0 is death. The primary purpose of its development was to allow physicians to evaluate a participant's ability to survive chemotherapy for cancer.
  participants
    90-100% = normal activity, few symptoms of disease | 58
    70-80% = normal activity, symptoms, cannot work | 25
    50-60% = needs help and needs medical care | 0
    <40% = disabled to severely disabled | 0
Number of Baseline Lesions (Target + Non-Target) by Independent Radiological Review [Number; unit: participants] — Target lesions are those measurable at baseline and are generally the largest lesions, most reliably measured and most representative of the participants sites of disease. Non target lesions are all of the sites of disease present at baseline not classified as target lesions. They include bone and cystic lesions and pleural/pericardial effusion/ascites. The Independent Reviewers only evaluated scans for those with baseline and follow-up scans.
  participants
    1 | 3
    2 | 6
    3 | 13
    4 | 10
    5 | 8
    >5 | 43

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Experiencing Treatment Emergent Adverse Events (TEAE)
Description: TEAEs were defined as adverse events (AEs) that began or worsened in severity on or after the date of the first dose of study drug and within 30 days of the last dose of study drug. A Serious AE (SAE) = any AE that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability, is a congenital anomaly/birth defect; constitutes an important medical event. Treatment-related AEs (TRAEs) were any TEAEs considered to be related to the study drug. A TRAE is a TEAE with relationship as suspected to either ABI-007 or gemcitabine The intensity of AEs were graded 1 to 5 according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. Other AEs not described in the CTCAE criteria, the intensity will be assessed by the investigator as mild grade (Gr 1), moderate (grade 2), severe (grade 3), life-threatening (grade 4) or death (grade 5)
Time Frame: Study drug initiation through 30 days after the last dose of study drug or End Of Study, whichever is later; maximum treatment duration was 54.9 weeks
Population: Safety population includes all enrolled participants who received at least 1 dose of study drug
Measure: Number; unit: participants
Groups:
- Nab-paclitaxel and Gemcitabine: Nab-paclitaxel 125 mg/m^2 by intravenous (IV) infusion over 30 - 40 minutes followed by gemcitabine 1000 mg/ m^2 IV infusion over 30 - 40 minutes once weekly for 3 weeks (Days 1, 8 and 15) followed by one week of rest (28 day cycle).
Arm/Group | Nab-paclitaxel and Gemcitabine
Number analyzed (Participants) | 83
participants
  At least 1 TEAE | 83
  At Least 1 Treatment-related TEAE | 82
  ≥ 1 TEAE with NCI CTCAE Gr 3 or higher | 70
  ≥ 1 TRAE NCI CTCAE ≥ Gr 3 | 62
  At Least 1 Serious TEAE | 20
  At Least 1 Treatment-related Serious TEAE | 9
  ≥ 1 TEAE causing discontinuing of either drug | 10
  ≥1 TRAE causing discontinuing of either drug | 5
  ≥ 1 TEAE causing reduction in ABI-007/Gemcitabine | 38
  ≥ 1 TRAE causing reduction in ABI-007/Gemcitabine | 38
  ≥1 TEAE causing interruption in either study drug | 43
  ≥1 TRAE causing interruption in either study drug | 40
  At Least 1 TEAE With Outcome of Death | 8
  ≥1 TRAE with Outcome of Death | 2

2. Primary Outcome: Overall Response Rate (ORR) Based on Independent Radiological Review (IRR)
Description: ORR was defined as the percentage of participants who achieve a complete response (CR) or partial response (PR) based on independent radiological review per Response Evaluation Criteria in Solid Tumors (RECIST) Criteria (V1.0). Using RECIST Version 1.0, participants were to achieve either a complete response defined as the disappearance of all known disease and no new sites or disease related symptoms confirmed at least 4 weeks after initial documentation or partial response defined as at least a 30% decrease in the sum of the longest diameters of target lesions and no progression in non-target lesions based on confirmed responses from the independent radiological review of best overall response during study treatment.
Time Frame: Assessment every 8 weeks; Day 1 to data cut off of 01 June 2015; Up to approximately 70 weeks
Population: Intent to Treat (ITT) population included all participants enrolled into the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nab-paclitaxel and Gemcitabine
Number analyzed (Participants) | 83
percentage of participants | 35 [24.8 to 46.2]

3. Secondary Outcome: Duration of Response (DoR) Based on IRR According to RECIST Guidelines
Description: DoR was defined as the time from the first tumor assessment when the confirmed CR/PR response criterion is met to the date of disease progression based on IRR following RECIST 1.0. Only for those participants with a confirmed CR/PR. If a participant had disease progression, then the date of disease progression was the event date. For a participant who did not develop disease progression or disease progression occurred after 2 or more missing tumor assessments, the participant was censored on the date of last tumor assessment where the participant was documented to be progression free. If a participant died prior to disease progression, the participant was censored on the date of death. If patient started new anti-cancer therapy, the patient was censored on the last tumor assessment date on or prior to the start date of new anti-cancer therapy
Time Frame: Assessment performed every 8 weeks; from the first participant enrolled to cut off date of 01 June 2015; up to approximately 70 weeks
Population: Includes participants with a Confirmed Complete or Partial Response
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Nab-paclitaxel With Gemcitabine: Nab-paclitaxel 125 mg/m^2 by intravenous (IV) infusion over 30 - 40 minutes followed by gemcitabine 1000 mg/ m^2 IV infusion over 30 - 40 minutes once weekly for 3 weeks (Days 1, 8 and 15) followed by one week of rest (28 day cycle).
Arm/Group | Nab-paclitaxel With Gemcitabine
Number analyzed (Participants) | 29
months | 8.9 [6.01 to 8.94]

4. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival (OS)
Description: Overall survival was defined as the time from the date of first treatment to the date of death. Participants who did not die at the end of study or clinical data cut were censored on the last-known-to-be-alive date or the clinical cut-off date, whichever was earlier.
Time Frame: From the first participant enrolled to data cut off of 01 June 2015; up to approximately 70 weeks
Population: ITT population includes all enrolled participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-paclitaxel With Gemcitabine
Number analyzed (Participants) | 83
months | 9.2 [7.60 to 11.10]

ADVERSE EVENTS:
Time Frame: TEAE that started: 1) From the date of first dose of study drug through 30 days after the last dose of study drug; collected from 20 Jan 2014 to 04 Aug 2016.
Description: 2) SAE's that had not resolved upon participants discontinuation were followed until recovered, recovered with sequelae, not recovered (death due to another cause) or death (due to the SAE); all AEs were assessed/monitored up to 132 weeks + 3 days
Arm/Group | Nab-paclitaxel and Gemcitabine
Serious Adverse Events (participants affected / at risk) | 22/83
Other Adverse Events (participants affected / at risk) | 83/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-paclitaxel and Gemcitabine (N=83)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 1
Local swelling (General disorders) | 1
Pyrexia (General disorders) | 2
Haemobilia (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Lymphangitis (Infections and infestations) | 1
Platelet count decreased (Investigations) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-paclitaxel and Gemcitabine (N=83)
Anaemia (Blood and lymphatic system disorders) | 26
Erythropenia (Blood and lymphatic system disorders) | 7
Leukopenia (Blood and lymphatic system disorders) | 56
Lymphopenia (Blood and lymphatic system disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 55
Thrombocytopenia (Blood and lymphatic system disorders) | 45
Abdominal distension (Gastrointestinal disorders) | 13
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 12
Ascites (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 23
Diarrhoea (Gastrointestinal disorders) | 17
Dyspepsia (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 41
Vomiting (Gastrointestinal disorders) | 33
Asthenia (General disorders) | 11
Chills (General disorders) | 5
Fatigue (General disorders) | 39
Oedema peripheral (General disorders) | 19
Pyrexia (General disorders) | 29
Hyperbilirubinaemia (Hepatobiliary disorders) | 12
Lung infection (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 7
Alanine aminotransferase increased (Investigations) | 22
Aspartate aminotransferase increased (Investigations) | 17
Blood alkaline phosphatase increased (Investigations) | 10
C-reactive protein increased (Investigations) | 7
Fibrin D dimer increased (Investigations) | 6
Gamma-glutamyltransferase increased (Investigations) | 11
Haemoglobin decreased (Investigations) | 50
Neutrophil count decreased (Investigations) | 7
Platelet count decreased (Investigations) | 11
Weight decreased (Investigations) | 7
White blood cell count decreased (Investigations) | 11
Decreased appetite (Metabolism and nutrition disorders) | 43
Hyperglycaemia (Metabolism and nutrition disorders) | 17
Hypoalbuminaemia (Metabolism and nutrition disorders) | 21
Hypocalcaemia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 15
Hyponatraemia (Metabolism and nutrition disorders) | 12
Hypoproteinaemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 5
Hypoaesthesia (Nervous system disorders) | 26
Neuritis (Nervous system disorders) | 6
Neuropathy peripheral (Nervous system disorders) | 10
Insomnia (Psychiatric disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 30
Nail disorder (Skin and subcutaneous tissue disorders) | 7
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 9
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present study data provided that the investigator shall (i) furnish the sponsor a copy of any proposed publication or presentation generally sixty (60) days in advance of the submission, (ii) delete any confidential information of the sponsor, and (iii) delay submission for generally up to ninety (90) days to permit the preparation and filing of intellectual property applications or until sponsor gives its consent in a timely manner